CLINICAL TRIAL: NCT06942468
Title: Efficacy and Safety of Topical Nano Preparation of Phenytoin Plus Fractional CO2 Laser Versus Fractional CO2 Laser Alone for Treatment of Atrophic Post Acne Scars: A Randomized Split Face Study.
Brief Title: Phenytoin in Treatment of Atrophic Post Acne Scars.
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohamed Abdalla Sultan, Dermatologist resident, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Phenytoin in post acne scars.
Record Dates: First submitted 2025-04-07; First posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Atrophic Acne Scar
MeSH Terms: interventions — Phenytoin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical Phenytoin and Fractional CO2 laser (Experimental): Topical Phenytoin and Fractional CO2 laser will be used in combinaton to treat atrophic post-acne scars.
  Interventions: Drug: Topical nano preparation of Phenytoin
- Fractional CO2 laser alone (Experimental): Fractional CO2 laser will be used alone to treat atrophic post acne scars.
  Interventions: Device: Fractional CO2 laser

INTERVENTIONS:
Drug: Topical nano preparation of Phenytoin — Topical nano preparation of Phenytoin will be used to treat atrophic post-acne scars. It will be in form of spanlastics.
  Other Names: Topical Phenytoin
  Arms: Topical Phenytoin and Fractional CO2 laser
Device: Fractional CO2 laser — Fractional CO2 laser will be used alone for treatment of atrophic post acne scars.
  Arms: Fractional CO2 laser alone

SUMMARY:
To evaluate the efficacy and safety of topical phenytoin spanlastics as an adjuvant therapy in treatment of atrophic post acne scars.

To compare the efficacy of topical phenytoin spanlastics combined with fractional co2 laser versus fractional co2 laser alone in treatment of atrophic post acne scars.

DETAILED DESCRIPTION:
Acne is one of the most dermatological problems in the world which causes scars as secondary damage .

It affects the appearance and psychology of the patient badly . There are three main types of scars: atrophic, hypertrophic, or keloidal depending on a loss (atophic) or gain (hypertrophic and keloidal) of collagen .

Atrophic scars presented in the form of icepick, rolling and poxscar . It is a challenge to mange atrophic scars because these scars result from tissue loss during the healing after severe acne. There are many therapeutic techniques that continuously evolving for management of these scars as: fractional lasers, microneedling, chemical peels and dermabrasion .

Phenytoin (PHT) is the main treatment for epilepsy. However, many patients who took it show gingival hyperplasia . Phenytoin causes increased fibroblasts proliferation. It has the ability to reduce the oedema and inflammation at the wound base and margins, early separation of slough, and collagen production and acceleration of growth of healthy granulation tissues, so it can be used in healing .

By induction of collagen synthesis and reducing inflammation, topical phenytoin can alleviate the appearance of atrophic scars including acne scars and improve their texture. Application of phenytoin directly to affected areas may lead to significant improvements in scarred skin over regular and consistent usage .

To the best of our knowledge, only one study has investigated the healing potential of PHT cream with microneedling application for the management of atrophic acne scars .

Nevertheless, its limited solubility, bioavailability, and inefficient distribution during topical administration limit its use. Nanopreparation of phenytoin showed promising findings that encourage the potential use of phenytoin loaded lipid nanoparticles for future topical application.

Spanlastics are composed of a non-ionic surfactant and an edge activator (EA). The presence of EA confers the penetration-enhancing effect of spanlastics that facilitate topical drug delivery. Spanlastics squeeze themselves through skin pores without being disrupted due to their elastic, deformable nature. Besides, spanlastics are non-immunogenic, biodegradable systems that are compatible with biological membrane with minimum toxicity. Given these premises of spanlastics as topical drug delivery systems, the current study is set to explore their features to enhance the penetration of phenytoin, control its release, and improve its efficacy in the management of atrophic acne scars.

Fractional carbon dioxide laser (CO2 laser) is the gold standard for the treatment of atrophic acne scars and skin rejuvenation . Its wavelength is 10,600nm. It targets water containing cells, which is its chromophore . It thermally acts on a portion of the skin creating numerous microthermal treatment zones leaving normal skin intact in between, which rapidly regenerates the ablated columns of tissue. Thermal injury induces coagulation and denaturation of collagen and reepithelialisation .

CO2 lasers have a double effect as they induce renewable processes of the wound and increase production of myofibroblasts and matrix proteins such as the hyaluronic acid.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged equal or more than 18 years old with atrophic post acne scars.

Exclusion Criteria:

* Pregnancy and lactation
* Hypertrophic scars
* Kidney, liver, neurological, haematological, malignant or immunosuppressive diseases.
* Active infection at the site of the scars
* Patients use medications that reduced tissue healing during the study or in a period less than one month ago (immunosuppressants and isotretinoin).

  * Patients who are taking anticoagulants or NSAIDS within the past 48h.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
To assess the Quantitative Global Acne Scarring score before. | Immediately at the end of the treatment and 2 months after the end of the treatment
  * The Quantitative Global Scarring Grading System uses a scale of 0 to 84
  * The scale assesses the severity of scarring based on the appearance, depth, and area of the scars.

REFERENCES:
- [Background] Sadeghzadeh-Bazargan A, Pashaei A, Ghassemi M, Dehghani A, Shafiei M, Goodarzi A. Evaluation and comparison of the efficacy and safety of the combination of topical phenytoin and microneedling with microneedling alone in the treatment of atrophic acne scars: A controlled blinded randomized clinical trial. Skin Res Technol. 2024 Jun;30(6):e13766. doi: 10.1111/srt.13766. PMID 38807440
- [Background] Rivera AE. Acne scarring: a review and current treatment modalities. J Am Acad Dermatol. 2008 Oct;59(4):659-76. doi: 10.1016/j.jaad.2008.05.029. Epub 2008 Jul 26. PMID 18662839